CLINICAL TRIAL: NCT06904508
Title: Electrophysiological Correlates of Anxiety-related Improvements Following Cognitive Behavioral Therapy for Autistic Youth in High-Need Communities
Brief Title: Brain Activity Changes After Cognitive Behavioral Therapy for Anxiety in Autistic Youth From High-Need Communities
Acronym: IAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montclair State University (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-FY23-24-3257; CDMRP-AR230226 (Other Grant/Funding Number: DoD Congressionally-Directed Medical Research Program)
Record Dates: First submitted 2025-02-21; First posted 2025-04-01 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder; Anxiety
Keywords: autism; autism spectrum disorder; anxiety; youth; randomized controlled trial; cognitive behavioral therapy; electroencephalogram
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist-Control Condition (No Intervention): Waitlist Control (WC) with Treatment-as-Usual (TAU). Participants in the WC arm will continue in their usual services and will be provided with referrals if needed. No specific treatment recommendations will be given.For ethical reasons, after completing the TAU waitlist period, families will be provided with an opportunity to participate in the FYF intervention.
- Treatment Condition: Facing Your Fears (FYF) Group (Experimental): The group consists of 4-6 families who will meet for 90-minute weekly sessions for 12-14 weeks. The sessions will focus on psychoeducation and implementing CBT techniques to help autistic youth and their caregivers "face their fears" and tackle their anxiety.
  Interventions: Behavioral: Facing Your Fears (FYF) Intervention: A CBT Focused Group Treatment for Autistic Youth with Anxiety

INTERVENTIONS:
Behavioral: Facing Your Fears (FYF) Intervention: A CBT Focused Group Treatment for Autistic Youth with Anxiety — FYF is an outpatient, multi-family, evidence-based CBT group treatment for children and adolescents ages 8-14 with average intellectual abilities, and a primary co-occurring anxiety diagnosis (social, generalized, separation anxiety, or specific phobia).
  Arms: Treatment Condition: Facing Your Fears (FYF) Group

SUMMARY:
The goal of this clinical trial is to investigate neural constructs related to anxiety symptoms in response to Facing Your Fears (FYF) treatment in autistic participants with co-occurring anxiety.

Researchers will compare participants receiving immediate FYF intervention to those in the waitlist control group (receiving treatment as usual) to see if there are differences in neural constructs and anxiety symptom changes over the study period.

Participants will:

* Complete the Facing Your Fears (FYF) intervention if assigned to the immediate treatment group
* Continue their usual treatment during a waitlist period if assigned to the control group, followed by the opportunity to participate in FYF intervention after the waiting period ends
* Complete assessments of neural constructs, anxiety symptoms, and other measures

DETAILED DESCRIPTION:
Aims of the study:

* How do brain activity patterns (measured by EEG) relate to anxiety symptoms in autistic youth, as reported by both the youth and their parents?
* Will brain activity changes line up with improvements in anxiety after FYF treatment in autistic youth from underserved communities?
* Will brain activity relate to other factors related to anxiety (e.g., a person's ability to handle uncertainty and manage emotions)?

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 8 and 14
* Have significant deficits in reciprocal social behavior as defined by a score of 11 or above on the parent-report SCQ questionnaire
* Are verbally fluent in English, enabling them to participate in the appropriate modules (3 or 4) of the researcher-administered ADOS-2
* Have an estimated verbal IQ of 70 or above as determined by the researcher-administered KBIT-2
* Have clinically significant anxiety symptoms as defined by significant elevations on either the parent-report SCARED questionnaire or the parent-report PRAS-ASD questionnaire
* Have a legal guardian who can provide consent for their child's participation as well as their own participation in the intervention alongside their child. If the legal guardian is unable to participate in the intervention themselves but would like for their child to receive the intervention with another caregiver who lives with the child, the legal guardian will still be the one to sign the consent form, but will provide permission for another caregiver (logged on the consent form) to participate in the intervention alongside the child

Exclusion Criteria:

* Fail to meet any of the above inclusion criteria
* If it is determined by the research team via parent report or direct observation that the child has a severe medical or psychiatric impairment (e.g., psychosis, severe aggressive behavior, or other severe clinical symptoms) that require more intensive treatment such as day treatment or hospitalization

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The Screen for Child Anxiety and Related Disorders (SCARED-P/C) | Baseline and within 2 weeks of intervention completion (up to 14 weeks post first intervention session)
  The Screen for Child Anxiety and Related Disorders - Parent/Child versions (SCARED-P/C) is comprised of five anxiety subscales, including panic, generalized anxiety, separation anxiety, and school avoidance symptoms, and a total anxiety subscale. The SCARED-P and SCARED-C each include 41 items designed to evaluate a child's recent anxiety symptoms. Participants rate their responses on a 3-point Likert scale: 0 (Not True or Hardly Ever True), 1 (Somewhat or Sometimes True), and 2 (Very True or Often True). A total score of 25 or higher is considered indicative of clinically significant anxiety. The SCARED has shown good psychometric properties across autistic and non-autistic samples. It has shown evidence for treatment sensitivity in previous FYF trials, and will be used as a primary outcome measure in this study as well.
Anxiety Scale for Children-Autism Spectrum Disorder Scale (ASC-ASD) | Baseline and within 2 weeks of intervention completion (up to 14 weeks post first intervention session)
  The Anxiety Scale for Children-Autism Spectrum Disorder Scale (ASC-ASD) is a self- and parent-report measure developed to assess separation anxiety, uncertainty, performance anxiety, and anxious arousal dimensionally in the autistic population. It consists of 25-items (scored 0-3) with higher scores indicating higher anxiety levels..
Parent Rated Anxiety Scale for Autism Spectrum Disorder (PRAS-ASD) | Baseline and within 2 weeks of intervention completion (up to 14 weeks post first intervention session)
  It consists of 25-items (scored 0-3) with higher scores indicating higher anxiety levels. This measure was developed to assess DSM-5 and anxiety symptoms distinct to ASD, specifically this measure takes the unique approach of examining behaviorally oriented anxiety symptoms. This measure has demonstrated reliability and validity in the autism population.
Error Related Negativity (ERN) Event-Related Potential (ERP) | Baseline and within 2 weeks of intervention completion (up to 14 weeks post first intervention session)
  EEG systems will be used to record Error Related Negativity using the Flanker paradigm. The Flanker paradigm involves congruent (50%) and incongruent (50%) trials with arrows facing the same direction as (congruent) or the opposite direction of (incongruent) the target. The order of congruent and incongruent trials will be random. All stimuli will be presented for 200 ms followed by an inter-trial interval that varies randomly from 2,300 to 2,800 ms. The participant will be given detailed task instructions, and receive feedback based on their performance at the end of each block. Error and correct trials will be separately averaged, with the error response as the mean activity between -25 and 75ms after the error response at scalp site where error-related brain activity is maximal. In addition, the correct response negativity (CRN) will be evaluated for the same time window and site on correct trials. The ERN (i.e., the error response minus CRN) will then be calculated for analysis
Electroencephalogram (EEG) Hemispheric Asymmetry | Baseline and within 2 weeks of intervention completion (up to 14 weeks post first intervention session)
  Resting EEG data will be collected for 6 minutes alternating between 1-min blocks of eyes open or closed (with the order counterbalanced across subjects). Baseline frontal alpha-band power during eyes-open rest will be calculated across the epoch using wavelet analysis for central frequencies (7.5-12.5 Hz) using 20 logarithmic steps at 7 cycles. To normalize the data, natural log-transformed scores will be calculated. Asymmetry scores were created as Ln(Left) - Ln(Right) for mean alpha power across F3(L)/4(R) and F7(L)/8(R) pairs.

SECONDARY OUTCOMES:
Child Behavior Checklist (CBCL) | within 2 weeks of intervention completion (up to 14 weeks post first intervention session)
  The Child Behavior Checklist is a 118-item parent-report measure that assesses broad psychopathology in children and adolescents. In this sample, the CBCL will be used to assess behavioral metrics related to anxiety. Parents rate each item on a 3-point scale (0-2). Raw scores are converted to t-scores, with elevated t-scores indicating behavioral or emotional problems.
Emotion Dysregulation Inventory (EDI) | within 2 weeks of intervention completion (up to 14 weeks post first intervention session)
  The Emotion Dysregulation Inventory is a 30-item parent-report questionnaire developed to assess facets of emotion dysregulation in autism spectrum disorder in the past seven days. These facets include reactivity (i.e., behavioral responses) and dysphoria (i.e., mental processes). Items are rated on a five-point scale (0-4) with higher ratings indicating greater dysregulation. The EDI contains two subscales: the reactivity (i.e., behavioral responses) and the dysphoria (i.e., mental processes) scale. The EDI has demonstrated both reliability and validity in the autism population.
Treatment Fidelity | Each intervention session (up to 14 weeks)
  Treatment Fidelity Measure assesses absence/presence of FYF treatment components; acceptability/usefulness of activities are rated. The measure utilizes a checklist format to assess the presence or absence of core treatment components on a session-by-session basis. In addition, a rating of quality will be assigned on a Likert scale ranging from poor (1), to adequate (3), to excellent (5) quality.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Kang, PhD, Principal Investigator — Montclair State University
Locations (2):
- United States (2):
  - Montclair State University, Montclair, New Jersey
  - Drexel University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
The study team will meet all results reporting requirements of the funding and regulatory agencies.